CLINICAL TRIAL: NCT01332812
Title: Dexamethasone for the Prevention of Postoperative Cognitive Dysfunction in Elderly Patients Undergoing to General Anesthesia
Brief Title: Dexamethasone for the Prevention of Postoperative Cognitive Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Duke University (Other)
Responsible Party: Principal Investigator, Maria José Carvalho Carmona, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Maria J.C. Carmona
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Dexamethasone; Postoperative cognitive dysfunction; General Anesthesia; neuropsychological tests
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Dexamethasone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone, POCD, psycological tests (Experimental): Subjects will be randomly assigned in two groups: For the Dexamethasone group, 8mg of dexamethasone will be administered intravenously before the induction of general anesthesia. For Control Group, no Dexamethasone will be administered.
  Tests for evaluation of quality of life, depressive symptoms and neuropsychological battery to assess general mental status, learning, attention, visuospatial perception, immediate memory, operational and executive skills and recall, including processing speed. This assessment will be applied before surgery, and 3, 7, 21, 90 and 180 days after surgery.
  Interventions: Drug: Dexamethasone
- Control, POCD, psycological tests (Sham Comparator): Subjects will be randomly assigned in two groups: For the Dexamethasone group, 8mg of dexamethasone will be administered intravenously before the induction of general anesthesia. For Control Group, no Dexamethasone will be administered.
  Tests for evaluation of quality of life, depressive symptoms and neuropsychological battery to assess general mental status, learning, attention, visuospatial perception, immediate memory, operational and executive skills and recall, including processing speed. This assessment will be applied before surgery, and 3, 7, 21, 90 and 180 days after surgery.
  Interventions: Other: control group

INTERVENTIONS:
Drug: Dexamethasone — a dose of 8 mg of dexamethasone will be administered intravenously before induction of general anesthesia
  Other Names: The Dexamethasone and Index Bispectral
  Arms: Dexamethasone, POCD, psycological tests
Other: control group — General anesthesia, without additional interventions
  Other Names: Index Bispectral and not received the Desamethasone
  Arms: Control, POCD, psycological tests

SUMMARY:
This study aims to evaluate the possible effect of dexamethasone on prevention of cognitive dysfunction in the postoperative period of elderly patients undergoing to surgery under general anesthesia.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction is related with the use of opioids in the postoperative period, lack of physical activity, fatigue, postoperative pain and quality of life. The use of corticosteroids preoperatively reduces postoperative pain, fatigue, nausea and vomiting in the postoperative period and is frequently used as an adjuvant in anesthesia. This study aims to evaluate the possible effect of dexamethasone on prevention of cognitive dysfunction in the postoperative period of elderly patients undergoing to surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients over 60 years,
* underwent surgery for inguinal hernia repair, Nissen procedure, cholecystectomy or other surgeries midsize under general anesthesia and hospital stay expected within 72 hours.

Exclusion Criteria:

* age less than 60 years,
* history of brain disease or dementia, other psychiatric disorders that affect cognition,
* lack of proficiency in Portuguese,
* use of corticosteroids or opioid preoperatively.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Score in neuropsycological tests. | 6 months.
  Tests for evaluation of quality of life, depressive symptoms and neuropsychological battery to assess general mental status, learning, attention, visuospatial perception, immediate memory, operational and executive skills and recall, including processing speed. This assessment will be applied before surgery, and 3, 7, 21, 90 and 180 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Maria José C Carmona, M.D., Principal Investigator — Faculty of Medicine of the University of Sao Paulo
Locations (1):
- General Hospital of the University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Valentin LS, Pereira VF, Pietrobon RS, Schmidt AP, Oses JP, Portela LV, Souza DO, Vissoci JR, Luz VF, Trintoni LM, Nielsen KC, Carmona MJ. Effects of Single Low Dose of Dexamethasone before Noncardiac and Nonneurologic Surgery and General Anesthesia on Postoperative Cognitive Dysfunction-A Phase III Double Blind, Randomized Clinical Trial. PLoS One. 2016 May 6;11(5):e0152308. doi: 10.1371/journal.pone.0152308. eCollection 2016. PMID 27152422